CLINICAL TRIAL: NCT06786026
Title: QL1706 Plus Nab-paclitaxel +/- Bevacizumab As 1L Treatment in Recurrent or Metastatic Triple-Negative Breast Cancer: a Non-randomized, Multicenter Phase II Study
Brief Title: QL1706 Plus Chemotherapy +/- Bevacizumab in 1L Treatment of R/mTNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief Physician, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-BC-IIT-004
Record Dates: First submitted 2024-10-09; First posted 2025-01-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: TNBC, Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Bevacizumab; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL1706 +nab-P (Other)
  Interventions: Drug: QL1706; Drug: Nab paclitaxel
- QL1706 +nab-P+bevacizumab. (Other)
  Interventions: Drug: bevacizumab; Drug: QL1706; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: bevacizumab — bevacizumab
  Arms: QL1706 +nab-P+bevacizumab.
Drug: QL1706 — Bispecific antibody (bsAB) targeting PD-1 and CLTA-4
Drug: Nab paclitaxel — albumin-bound paclitaxel

SUMMARY:
This study is to evaluate the efficacy and safety of QL1706 plus albumin-bound paclitaxel ± bevacizumab in 1L treatment of r/mTNBC

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study and sign the informed consent form;
2. Female patients aged ≥18 years and ≤70 years old who had been dignosed with breast cancer;
3. According to the definition of the latest ASCO/CAP guidelines, histologically confirmed estrogen receptor negative (ER-) and progesterone receptor negative (PR-), human epidermal growth factor receptor 2 negative
4. For patients with locally advanced, recurrent or metastatic breast cancer who have not used any systematic treatment (it is allowed to accept adjuvant/neoadjuvant treatment, and the time from the last administration to recurrence and metastasis should be ≥ 6 months);
5. According to RECIST 1.1, there is at least one measurable lesion;
6. ECOG score: 0~1;
7. Tumor tissue specimens that can be used for biomarker detection;
8. Adequate organ function (no blood components or cell growth factor drugs are allowed within 14 days before the first medication): (1) Absolute neutrophil count ≥1.5×109/L; (2) Platelets ≥100×109/L; (3) Hemoglobin ≥90 g/L; (4) Serum albumin ≥30 g/L; (5) Thyroid-stimulating hormone (TSH) ≤1×ULN (if abnormal, the FT3 and FT4 levels should be examined at the same time. If the FT3 and FT4 levels are normal, you can be included in the group); (6) Serum total bilirubin ≤1.5×ULN，if liver metastasis is present, ≤3ULN; (7) ALT and AST ≤2.5×ULN, if liver metastasis is present, ALT and AST ≤5ULN; (8) AKP≤2.5×ULN; Serum creatinine ≤1.5×ULN; (9) International normalized ratio (INR) ≤1.5 (not receiving anticoagulant therapy).

Exclusion Criteria:

* 1.The presence of any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism;Those who suffer from vitiligo or whose asthma has been completely relieved in childhood and do not need any intervention in adulthood can be included; asthma that requires medical intervention with bronchodilators cannot be included); 2.Are currently using immunosuppressants or systemic steroid therapy to achieve immunosuppression ((in dosing exceeding 10 mg daily of prednisone equivalent), and are still using it within 2 weeks before enrollment; 3.Severe allergic reactions to other monoclonal antibodies; 4. Known history or evidence of interstitial lung disease or active non-infectious pneumonia; 5.Known central nervous system metastasis; 6.Known additional malignant tumors within the past 5 years (except cured basal cell carcinoma of the skin and cervical cancer in situ); 7. The presence of uncontrolled hypertension (systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg) or dignosis with hypertensive crisis or hypertensive encephalopathy. Known history of hypertension are admitted to the study if their blood pressure is controlled below this standard and maintained with antihypertensive therapy.

  8.Patients with a history of severe cardiovascular and cerebrovascular disease, including but not limited to: (1) NYHA grade 2 or above heart failure (2) Unstable angina (3) Myocardial infarction within 1 year (4) Clinically significant supraventricular infarction or ventricular arrhythmia requiring treatment or intervention (5) QTc>450ms (male); QTc>470ms (female); 9.Those who are receiving thrombolysis or anticoagulation therapy; prophylactically use of low-dose aspirin and low-molecular-weight heparin are allowed; 10.Have clinically significant bleeding symptoms or a clear bleeding tendency within 3 months before enrollment; if fecal occult blood is positive in the screening, it should be re-examined. If it is still positive after the reexamination, a gastroscopy is required; 11.The tumor invades vital blood vessels, or a high possibility that the cancer will invade important blood vessels in the future study period, which may lead to fatal bleeding; 12.Patients with pleural effusion, ascites or pericardial effusion that require drainage can be enrolled if the researcher assesses that the symptoms are stable after drainage; 13.Arterial/venous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; 14.Major vascular disease (for example, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months before the start of study treatment; 15.Urine routine shows urine protein ≥ ++ and confirmed 24-hour urine protein amount &gt;1.0 g; 16.Suffering from active infection, unexplained fever ≥38.5℃ within 7 days before taking the drug, or baseline white blood cell count &gt;15×109/L; 17.Those with congenital or acquired immune deficiency (such as HIV infection); those who are hepatitis B surface antigen (HBsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 2000 IU/ml, or hepatitis C virus antibody positive; Have received live vaccines less than 4 weeks before study medication or may be vaccinated during the study period; 18.In the judgment of the researcher, the patient has other factors that may affect the study results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) that require combined treatment, and serious laboratory tests. Abnormalities, accompanied by family or social factors, may affect the patient&#39;s safety.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator | At baseline, at the time point of every 6 weeks, up to 1 years
  ORR (Objective response rate) is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response) or PR (partial response) per RECIST v1.1.

SECONDARY OUTCOMES:
DCR by investigator | At baseline, at the time point of every 6 weeks, up to 1 year
  DCR (Disease control rate) is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response), PR (partial response) or SD (stable disease) per RECIST v1.1.
Safety (incidence rate of adverse event) | From time of informed consent provided to 3 months after the last dose of study therapy
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. Percentage of participants who experienced an adverse event and discontinued study drug due to an AE.
PFS (Progression-Free Survival) | Up to 2 years
  PFS is the time from the date of the first dose until the date of documented radiographic disease progression or death (by any cause in the absence of progression).
OS (Overall Survival) | Up to 3 years
  OS is the time from the date of the first dose until the date of death by any cause.

OTHER OUTCOMES:
Exploratory purposes | Up to 3 years
  The correlation between biomarkers such as PD-L1 subtype, Fudan subtype, HIM subtype, immune microenvironment subtype, and therapeutic efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No